CLINICAL TRIAL: NCT01133756
Title: An Open-Label, Multicenter, Randomized, Phase Ib/II Study of E7080 in Combination With Carboplatin + Gemcitabine Versus Carboplatin + Gemcitabine Alone as Second Line Therapy in Patients With Platinum-Sensitive Recurrent Ovarian Cancer by CA125.
Brief Title: E7080 in Combination With Carboplatin + Gemcitabine Versus Carboplatin + Gemcitabine Alone as Second Line Therapy in Patients With Platinum-Sensitive Recurrent Ovarian Cancer by CA125
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Eisai Inc. (Industry)
Collaborators: PharmaBio Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-701; 2009-016050-41 (EudraCT Number)
Record Dates: First submitted 2010-05-21; First posted 2010-05-31 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2016-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — lenvatinib; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lenvatinib plus carboplatin + gemcitabine (Experimental): Phase IB and Phase II
  Interventions: Drug: Lenvatinib; Drug: Carboplatin; Drug: Gemcitabine
- Carboplatin + gemcitabine (Active Comparator): Phase II
  Interventions: Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Lenvatinib — lenvatinib (as 1mg, 4mg, and 10mg tablets) was administered orally, once daily continuously for each 21-day treatment cycle.
  Other Names: Lenvima, E7080
  Arms: Lenvatinib plus carboplatin + gemcitabine
Drug: Carboplatin — Carboplatin was to be administered on Day 1 of every 21-day cycle at a dose AUC 4 over 30 minutes.
Drug: Gemcitabine — Gemcitabine was to be administered on Day 1 and Day 8 of every 21-day cycle at a dose of 1000 mg/m2 over 30 minutes.

SUMMARY:
The purpose of this study was to determine the maximum tolerated dose (MTD)/recommended Phase II dose of lenvatinib administered in combination with carboplatin and gemcitabine (Phase IB) and to evaluate the safety and tolerability of E7080 administered in combination with carboplatin and gemcitabine compared to carboplatin and gemcitabine alone (Phase II) in participants with platinum-sensitive recurrent ovarian cancer.

DETAILED DESCRIPTION:
This open-label, multicenter, randomized study was to consist of a Phase 1b portion: a safety run-in period with 3 doses of lenvatinib administered in combination with carboplatin + gemcitabine; and a Phase II portion: a randomized 2-arm period. Approximately 100 participants with ovarian cancer were to be enrolled in the study (10 to 20 participants in the Phase 1b portion and 80 participants in the Phase II portion). Participants were to participate in either the Phase 1b or the Phase II portion. Participants were to receive study treatment (lenvatinib plus carboplatin + gemcitabine or carboplatin + gemcitabine) for six 21-day cycles (18 weeks). Participants who receive E7080 and experience evidence of clinical benefit (CR, PR, or SD) may continue single agent E7080 beyond 18 weeks, until the occurrence of progressive disease (PD), unacceptable toxicity, withdrawal of consent, or withdrawal by investigator, whichever occurs first.

Initially, an ascending dose schedule starting at lenvatinib 16 mg once daily on Day 1 to Day 21 was chosen for the Phase 1b portion to determine the MTD of lenvatinib administered once daily in combination with carboplatin + gemcitabine; however, due to hematologic toxicity observed in the first cohort, the lenvatinib administration schedule was changed to Days 2 to 21 in Protocol Amendment 2. Continued hematologic toxicity prompted a third protocol amendment, designed to evaluate a lower range of doses starting at lenvatinib 8 mg once daily in Protocol Amendment 3.

After three protocol amendments, recruitment into the Phase 1b portion of the study was very limited, with only one evaluable participant enrolled during the last 5 months of recruitment. Due to the limited enrollment despite significant diligence to boost enrollment and the complex study design required to manage hematologic toxicity, the study was terminated before the initiation of Phase II.

Safety was assessed by the monitoring and recording of all adverse events (AEs) and serious adverse events (SAEs); vital signs; Gynecological Oncology Group performance status; clinical laboratory evaluations; physical examinations; and 12-lead electrocardiograms (ECGs).

ELIGIBILITY:
Inclusion Criteria:

Participants may be in the study only if they meet all of the following criteria.

1. Female participants greater than or equal to 18 years of age.
2. Histologically or cytologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer that was treated with and was sensitive to one prior platinum-based chemotherapy regimen for Stage III or Stage IV disease.
3. Documentation of biochemical relapse defined by CA125 criteria (measurable or non-measurable by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST criteria), more than six months since completion of first-line platinum-based chemotherapy requiring treatment with further platinum-based chemotherapy. CA125 criteria for relapse Gynecologic Cancer Intergroup (GCIG) criteria are the finding of 2 serum CA125 levels with samples taken at least 1 week apart and no greater than 3 months apart:

   1. greater than or equal to 2 x ULN in participants with an elevated pre-treatment serum CA125 level followed by normalization on treatment and prior to progression OR
   2. greater than or equal to 2 X nadir value for participants with an elevated pre-treatment CA125 that never normalizes).
4. Gynecological Oncology Group performance status of 0 or 1
5. Life expectancy greater than or equal to 3 months
6. Participants must have recovered from effects of any major surgery within 28 days from the first dose of study treatment.
7. Adequate hematologic, renal, liver, and coagulation system function as defined by laboratory values performed within 21 days prior to initiation of dosing.

   1. Absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L
   2. Platelet count greater than or equal to 100 x 109/L
   3. Hemoglobin greater than or equal to 9 g/dL
   4. Serum creatinine less than or equal to 1.5 X ULN and/or creatinine clearance 50 dL/min
   5. Total serum bilirubin less than or equal to 1.5 X ULN
   6. Serum aspartate transaminase (AST/SGOT) or serum alanine transaminase (ALT/SGPT) less than or equal to 2.5 X ULN, and less than or equal to 5 X ULN in cases of liver metastasis
   7. PT/International normalized ratio (INR) less than or equal to 1.5 X ULN
   8. h. PTT less than or equal to 1.1 X ULN
8. Blood pressure must be well-controlled (less than or equal to 140/90 mmHg at screening) with or without antihypertensive medication. Participants must have no history of hypertensive crisis or hypertensive encephalopathy;
9. Participants should have a negative pregnancy test at screening in pre-menopausal women and women less than 2 years after the onset of menopause. Pre-menopausal women must agree to use an acceptable method of birth control from the time of the negative pregnancy test up to 90 days after the last dose of study drug. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for greater than or equal to 1 year;
10. Before study entry, written informed consent must be obtained from participant prior to performing any study-related procedures.

Exclusion Criteria:

Participants will not be entered in the study for any of the following reasons:

1. Pregnant, breast-feeding, or refusing double barrier contraception, oral contraceptives or avoidance of pregnancy measures;
2. Prior anti-angiogenic therapy with anti-VEGFR inhibitors; bevacizumab is allowed;
3. Prior gemcitabine;
4. Participants with proteinuria greater than 1+ on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with 24-hour urine protein greater than or equal to 1 g/24 hours will be ineligible.
5. Ovarian nonepithelial cancer, including malignant mixed Mullerian tumors and borderline tumors (e.g., tumors of low malignant potential);
6. Other malignancy within 5 years of randomization, with the exception of adequately treated carcinoma in situ of the cervix or non-melanoma skin cancer, with no subsequent evidence of recurrence;
7. History of, or known carcinomatous meningitis;
8. Are currently receiving any other treatment for the tumor (including palliative radiotherapy) aside from control of symptoms;
9. Received treatment in another clinical study within the 30 days prior to commencing study treatment or participants who have not recovered from side effects of an investigational drug to Grade less than or equal to 1, except for peripheral neuropathy (Grade 1 or 2 are permitted) or alopecia;
10. Received chemotherapy, biological therapy, hormonal therapy, targeted therapy, or radiotherapy within the 30 days prior to commencing study treatment or have not recovered from all treatment-related toxicities to Grade less than or equal to 1, except for peripheral neuropathy (Grade 1 or 2 are permitted) or alopecia;
11. Serious non-healing wound, ulcer, bone fracture, or have undergone a major surgical procedure, open biopsy, or significant traumatic injury within the 28 days prior to commencing study treatment. Minor surgery such as Portacath placement or skin biopsy is permitted if greater than or equal to 7 days have passed;
12. The use of anti-coagulants such as Vitamin K antagonists, unfractionated heparin, or low molecular weight heparin;
13. Refractory nausea and vomiting, malabsorption, significant bowel resection, or any other medical condition that would preclude adequate absorption or result in the inability to take oral medication;
14. Significant cardiovascular impairment (history of congestive heart failure) New York Heart Association (NYHA) Grade II, unstable angina or myocardial infarction within the past 6 months, or serious cardiac arrhythmia);
15. Any history of cerebral vascular accident (CVA) or transient ischemic attack (TIA) unless they have had no evidence of active disease for at least 6 months prior to randomization
16. Active hemoptysis (defined as bright red blood of 1/2 teaspoon or more) within the 30 days prior to study entry;
17. History of abdominal fistula, gastrointestinal perforation, or intrabdominal abscess within the 6 months prior to enrolment;
18. History of bleeding diathesis or coagulopathy;
19. History of an allograft requiring immunosuppression;
20. Known positive human immunodeficiency virus (HIV), known surface antigen positive for hepatitis B hepatitis or C positive;
21. Hypersensitivity to E7080 and/or E7080 chemical derivative; or
22. Have any other uncontrolled infection or medical condition which would interfere with the conduct of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harish Dave, MD, Study Director — Quintiles, Inc.
Locations (1):
- Texas Oncology - Austin Central, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Approximately, 100 participants were planned to be enrolled (10-20 in Phase 1b and 80 in Phase 2) but only 7 participants were enrolled.
Groups:
- Lenvatinib 16 mg (Day 1 to Day 21) + Carboplatin + Gemcitabine: Participants received carboplatin (area under the concentration-time curve [AUC] 4) + gemcitabine (1000 mg/m2) intravenous (IV) infusion over 30 minutes in combination with lenvatinib 16 mg on Day 1 of 21-day cycle and gemcitabine (1000 mg/m2) alone on Day 8 of the cycle.
- Lenvatinib 16 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine: Participants received carboplatin (AUC 4) + gemcitabine (1000 mg/m2) IV infusion over 30 minutes in combination with lenvatinib 16 mg on Day 2 of 21-day cycle and gemcitabine (1000 mg/m2) alone on Day 8 of the cycle.
- Lenvatinib 8 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine: Participants received carboplatin (AUC 4) + gemcitabine (1000 mg/m2) IV infusion over 30 minutes in combination with lenvatinib 8 mg on Day 2 of 21-day cycle and gemcitabine (1000 mg/m2) alone on Day 8 of the cycle.
Period: Overall Study
Arm/Group | Lenvatinib 16 mg (Day 1 to Day 21) + Carboplatin + Gemcitabine | Lenvatinib 16 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine | Lenvatinib 8 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine
Started | 2 | 3 | 2
Completed 6 Cycles | 1 (One participant completed 6 cycles and remained in the study until 18 Sep 2012.) | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 2 | 3 | 2
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Investigator Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Progression of Disease | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lenvatinib 16 mg (Day 1 to Day 21) + Carboplatin + Gemcitabine: Participants received carboplatin (AUC 4) + gemcitabine (1000 mg/m2) IV infusion over 30 minutes in combination with lenvatinib 16 mg on Day 1 of 21-day cycle and gemcitabine (1000 mg/m2) alone on Day 8 of the cycle.
- Total: Total of all reporting groups
Arm/Group | Lenvatinib 16 mg (Day 1 to Day 21) + Carboplatin + Gemcitabine | Lenvatinib 16 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine | Lenvatinib 8 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine | Total
Number analyzed (Participants) | 2 | 3 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 2 | 3 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLTs were defined as clinically significant adverse events occurring less than or equal to 21 days after commencing study treatment and considered to be possibly or probably related to study treatment by the Investigator. If 1 DLT occurred at any dose level, the cohort was to be expanded to include a maximum of six evaluable subjects. If 2 DLTs occurred at any dose level, the maximum tolerated dose (MTD) was to be either defined as the preceding dose, or an intermediate dose. To evaluate an intermediate dose, an additional dose cohort could be added to more accurately define the MTD.
Time Frame: Cycle 1 (21 days)
Population: Safety analysis was evaluated based on Safety Population, defined as all subjects enrolled into the Phase 1b portion of this study, except for those who (i) dropped out of the study prior to receiving any study drug, or (ii) were without any safety assessments following the first dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Lenvatinib 16 mg (Day 1 to Day 21) + Carboplatin + Gemcitabine | Lenvatinib 16 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine | Lenvatinib 8 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine
Number analyzed (Participants) | 2 | 3 | 2
Participants
  Platelet count decreased | 1 | 0 | 0
  Thrombocytopenia | 0 | 2 | 0

2. Secondary Outcome: Biomarker CA125-based Overall Response Rate (B-ORR), Within Treatment Group
Description: Due to the limited enrollment despite significant diligence to boost enrollment and the complex study design required to manage hematologic toxicity, the study was terminated before the initiation of Phase 2. Hence the analysis was not conducted.
Time Frame: Day 1 of every cycle, at end of treatment visit and every 2 months during follow-up period for patients who complete study without progressive disease.
Population: Due to the limited enrollment despite significant diligence to boost enrollment and the complex study design required to manage hematologic toxicity, the study was terminated before the initiation of Phase 2. Hence the analysis was not conducted.
Arm/Group | Lenvatinib 16 mg (Day 1 to Day 21) + Carboplatin + Gemcitabine | Lenvatinib 16 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine | Lenvatinib 8 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Biomarker-based Proportion of Biomarker-Progression-Free Survival (B-PFS) at Week 12, Within Treatment Group
Description: as for outcome 2
Time Frame: Week 12
Population: as for outcome 2
Arm/Group | Lenvatinib 16 mg (Day 1 to Day 21) + Carboplatin + Gemcitabine | Lenvatinib 16 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine | Lenvatinib 8 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For each participant, from the first dose till 30 days after the last dose or up to 18 Sep 2012 or up to 2.5 years
Description: Treatment emergent adverse events (defined as an adverse event (serious or non-serious) that started/increased in severity on/after the first dose of study medication up to 30 days after the final dose of study medication) are reported.
Groups:
- Lenvatinib 8 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine: Participants received carboplatin (AUC 4) + gemcitabine (1000 mg/m2) intravenous (IV) infusion over 30 minutes in combination with lenvatinib 8 mg on Day 2 of 21-day cycle and gemcitabine (1000 mg/m2) alone on Day 8 of the cycle.
Arm/Group | Lenvatinib 16 mg (Day 1 to Day 21) + Carboplatin + Gemcitabine | Lenvatinib 16 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine | Lenvatinib 8 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/3 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 16 mg (Day 1 to Day 21) + Carboplatin + Gemcitabine (N=2) | Lenvatinib 16 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine (N=3) | Lenvatinib 8 mg (Day 2 to Day 21) + Carboplatin + Gemcitabine (N=2)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 2 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 2 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 2 | 1
BRADYCARDIA (Cardiac disorders) | 0 | 1 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 1
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 1 | 0 | 0
LIP SWELLING (Gastrointestinal disorders) | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1 | 0
ORAL DISORDER (Gastrointestinal disorders) | 0 | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 0 | 1
CHEST PAIN (General disorders) | 1 | 0 | 0
FATIGUE (General disorders) | 1 | 2 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 0 | 0
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 1
ABSCESS NECK (Infections and infestations) | 1 | 0 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 1 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 0 | 0
BLOOD ALBUMIN DECREASED (Investigations) | 1 | 0 | 0
BLOOD MAGNESIUM DECREASED (Investigations) | 1 | 0 | 0
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0 | 0
HAEMATOCRIT DECREASED (Investigations) | 1 | 0 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 1 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0
TREMOR (Nervous system disorders) | 1 | 0 | 0
PROTEINURIA (Renal and urinary disorders) | 1 | 1 | 0
BREAST MASS (Reproductive system and breast disorders) | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
SKIN ATROPHY (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
SWELLING FACE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 2 | 0
THROMBOSIS (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the limited enrollment despite significant diligence to boost enrollment and the complex study design required to manage hematologic toxicity, the study was terminated before the initiation of Phase 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other